CLINICAL TRIAL: NCT04509427
Title: Comparison of Video-based and Paper Instructional Material to Promote EXercise and Posture in Individuals with and Osteoporosis
Brief Title: Exercise and Posture in Individuals with Osteoporosis
Acronym: EXPO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not receive the human or monetary resources to get this study off the ground.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Donald Lein, Associate Professor, Director of Continuing Education and Community Outreach, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXPO OP TRIAL
Record Dates: First submitted 2020-06-29; First posted 2020-08-12 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis
Keywords: Exercise Training; Posture training; Web-based video instruction; Handouts
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: After baseline measurements, participants will be assigned to one of two groups. Both groups will receive the same intervention except one group will also receive video instruction of the program intervention. Both groups will receive intervention instruction handouts and video-conferencing with a physical therapist, who will provide initial instruction of the program, assist with program progression, and assess safety and quality of performance of the program by the participants.
Who Masked: Investigator
Masking Description: The physical therapist responsible for baseline and post-intervention measurements will not know group assignments of the participants. Participants will be told not to tell this physical therapist their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Handouts Only (HO) group (Active Comparator): The HO only group will receive program instructions via handouts and videoconferencing with a physical therapist who will provide intervention instruction, assist with program progression, and monitor participant quality of movement and safety.
  Interventions: Behavioral: Instructional handouts; Behavioral: Physical therapist instruction and monitoring via teleconferencing; Behavioral: Posture training; Behavioral: Marching in place
- Handouts plus web-based video (HO+) group (Active Comparator): The HO+ group will receive the same intervention as the HO group but they will also have access to web-based videos that will lead them through all exercise/posture routines like a commercial exercise video.
  Interventions: Behavioral: Instructional handouts; Behavioral: Physical therapist instruction and monitoring via teleconferencing; Behavioral: Web-based instructional videos; Behavioral: Posture training; Behavioral: Marching in place

INTERVENTIONS:
Behavioral: Instructional handouts — Handouts will include written instructions for each aspect of the multifaceted exercise/posture training program
Behavioral: Physical therapist instruction and monitoring via teleconferencing — The intervention physical therapist (PT) meets with them via Zoom for 60 minutes to help them start the program in the first week. This PT will meet with them again in week 2 to complete initial instructions. The PT will meet with them week 3 and then every other week for 15-minutes to help individuals safely progress the program.
Behavioral: Web-based instructional videos — Instructional videos that will lead participants through every part of the intervention - like a commercial exercise video.
  Arms: Handouts plus web-based video (HO+) group
Behavioral: Posture training — Participants will learn how to hold a neutral spine posture during sitting, forward leaning in sitting, sit-to-stand-to-sit, standing, forward leaning in standing, supine-to-sit-to-supine, supine-to-prone-to-supine, and lifting. Principles learned with these functional movement patterns will then be put to practice in common tasks like sweeping, washing dishes, dusting, and gardening. This will be taught over two sessions in the first two weeks of the program. To reinforce holding neutral spine with all activities, participants will perform a 5-minute posture warm-up routine prior to exercising.
Behavioral: Marching in place — Participants will perform marching in place five times a week. Participants will be instructed to slowly progress to a goal of performing 30 minutes of marching in place per session. They will be instructed to lift their knees to a height that is between their waist and knee when marching. They will be instructed to march between a rating of 10 -14 on the 20-point Borg scale for rate of perceived exertion

SUMMARY:
Osteoporosis is a common condition found in postmenopausal women. Osteoporosis increases the risk of fractures: especially hip and vertebral fractures. These fractures increase the risk of morbidity and mortality. Falls and movements that incorporate trunk flexion or rotation can increase the risk of fractures in women with osteoporosis. Weight-bearing exercise and posture training are important complementary therapies to help decrease the risk of fractures and improve the function of individuals with osteoporosis. Often in Rheumatology clinic, patient's will be given handouts concerning bone building exercises and tips on holding safe postures with activities to complete, with little follow-up of their progress or evaluation of their technique. In this study, we will compare a video-based exercise intervention with printed handout group to a handout only group and will evaluate the effectiveness of these two different modalities using physical activity measures and overall outcomes of strength and posture.

DETAILED DESCRIPTION:
Osteoporosis is a common condition found in postmenopausal women. Osteoporosis increases the risk of fractures: especially hip and vertebral fractures. These fractures increase the risk of morbidity and mortality. Falls and movements that incorporate trunk flexion or rotation can increase the risk of fractures in women with osteoporosis. Weight-bearing exercise and posture training are important adjunctive therapies to help decrease the risk of fractures and improve the function of individuals with osteoporosis. Often in Rheumatology and osteoporosis clinics, participant's will be given handouts concerning posture and exercise to complete, with little follow-up of their progress or evaluation of their technique. In this study, investigators will determine if the addition a video-based exercise intervention with handouts and limited physical therapist instruction and monitoring help this population increase adoption of a regular exercise program designed to improve lower extremity strength and dynamic posture.

The purpose of this study is to determine if the addition of computer-based video instructions with handouts and limited physical therapist (PT) instruction helps adoption and performance of an intervention designed to improve strength, dynamic posture, and balance in individuals with osteoporosis (OP). Investigators will perform all measurements and interventions via web-based and telecommunication technology. Twenty-four participants will be recruited for this feasibility study using flyers posted in the Rheumatology and Osteoporosis clinics at the University of Alabama at Birmingham (UAB). The investigators, who help staff these clinics, will also alert other clinic physicians of this study via flyers designed for these health care professionals to help recruit study participants. The participants will consent to participate in this study. The UAB Institutional Review Board will approve this study.

After consenting, a physical therapist (PT), blind to group assignment, will perform outcome measurements. Outcome measurements will be assessed at baseline and within a week after the 12-week intervention is completed. Measurements include five-time sit-to-stand-to sit (5xSTS), 4-stage balance test, and a dynamic posture test. Participants will also complete a questionnaire that examines demographics, medical history, exercise and fall perceptions, and functional activity performance. The pre- and post-intervention questionnaires will be similar except the post-intervention questionnaire will not include demographic, medical history questions, and perceived readiness to exercise item. SurveyMonkey will be used to deliver and collect all questionnaire data. The post-intervention questionnaire will contain items assessing intervention satisfaction.

Prior to enrolling participants, investigators will develop a script and checklist for the PT performing the measurements to increase consistency of outcome measurement. The PT will also practice these measurements using Zoom and intra-rater reliability will be determined. Intra-rater reliability will also be assessed from the data collected. Finally, investigators will perform quality control by reviewing recordings of the measurement sessions.

After baseline measurements, participants will be randomly assigned to one of two groups: one group will receive handouts that provide program instructions with PT coaching (HO) or a group who receives the same instructional delivery plus links to web-based videos instructing all elements of the program intervention (HO+). Participants will be asked to perform moderate level exercise/posture activity 5 sessions/week for 35 to 40 minutes per day (duration of activity/session by the end of the intervention). By email, the HO+ group participants will receive handouts with links to access the safe exercise posture instruction, posture warm-up, balance exercise resistance exercise and marching. The HO group will also receive an email that with the same attachments minus the video links. In both groups, the first intervention instruction email will instruct the participants to not start the program until the intervention PT (not the same PT who performs the measurements) guides them through the program via a Zoom videoconference. In week two, the intervention PT will finish the initial instructions in another 60-minute session. The PT will meet with participants during the third week of the intervention for a 15-minute meeting and will continue to meet with participants for 15-minutes every two weeks thereafter via Zoom. During these 15-minute sessions, the intervention PT will help individuals progress exercises, monitor symptoms, answer questions, and make performance recommendations. All participants will be instructed to track their posture and exercise activity by using a monitoring log provided by the research group. These logs will be shared with the investigators.

Both groups will perform marching in place five times a week. Participants will be instructed to slowly progress to a goal of performing 30 minutes of marching in place per session. They will be instructed to lift their knees to a height that is between their waist and knee when marching. Participants will start performing at 5 minutes of marching twice a day. Every two weeks they will progress the goal of marching time by 5 minutes. They will march two times per day until they reach 20 minutes. At this time, they will march one time per day. They will be instructed to march between a rating of 10 -14 on the 20-point Borg scale for rate of perceived exertion. The intervention PT will help participants in both groups progress safely when she teleconferences with each participant every two weeks.

Posture training will be performed daily. The participants will be taught how to hold good posture with activity over two 60-minute sessions by the intervention PT. In the first visit, the intervention PT will discuss holding dynamic posture basics, finding and holding good posture in sitting and sit to stand. In the next visit, she will teach them how to progress to standing activities while holding good posture. The PT will instruct the participant to use the posture activities as a warm-up on all days of exercise. She will also encourage participants to incorporate these skills in daily activities.

The intervention PT will use scripts and checklists developed prior to participant enrollment to ensure consistency of instruction between participants. The intervention PT will practice instructing participants prior to participant enrollment via Zoom with other investigators. These sessions will be taped so that they can be reviewed and scripts and checklists refined.

Demographic, satisfaction data, perception items and scales will be analyzed using appropriate descriptive statistics. Descriptive statistics, such as means and standard deviations, will also be used to describe data from 5xSTS and balance tests. These tests will also be analyzed using Cohen d to determine effect size. To determine within and between group differences over time, mixed-factor ANOVAs will be used. Finally, a Wilcoxon-Signed Rank test will be used to determine differences between the groups for the dynamic posture test.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females
* Age >50
* Confirmed Osteoporosis diagnosis by dual energy X-ray absorptiometryscan
* Ambulatory
* Able to read and speak English
* With access to a computer and/or smartphone to view video material

Exclusion Criteria:

* Currently meeting the recommended Physical Activity Guidelines for Americans
* Diagnosis of fibromyalgia or other chronic pain syndrome
* Any history of serious cardiac comorbidities or arrhythmias
* Any history of chronic pulmonary condition
* Any history of active cancer
* Any history of active venous thromboemblism
* Any bleeding disorder
* Currently undergoing a PT program or recently completed PT treatment within the last 12 weeks
* Any current orthopedic condition that would preclude patient from exercising regularly
* Any patient scheduled for a future surgical procedure
* Current chronic steroid therapy >10mg

Min Age: 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Change in 5 times sit to stand from baseline to 3 months | This test will be performed at baseline and within a week after the completion of the intervention
  5 times sit to stand is a test performed in clinic that assesses lower extremity strength and function. Using a stop watch, an investigator will record the time (in seconds) it takes for an individual to complete five sit-to-stand-to-sit cycles. The participants will cross their arms over their chest and will perform this test using a kitchen or dining room chair placed against the wall.

SECONDARY OUTCOMES:
Change in the 4-stage balance test from baseline to 3 months | This test will be performed at baseline and within a week after the completion of the intervention.
  This is a balance test that consists of four positions: stand with feet together, modified tandem stance, tandem stance, and standing on one foot. Participants will perform these tests standing by a wall to allow them to catch themselves if they lose their balance. All participants will start with feet together. They will hold this position for 10 seconds. If successful, they will progress to holding a modified tandem position for 10 seconds. The next position is tandem stance and then finally standing on one foot if they can hold tandem stance for 10 seconds. For the modified tandem stance and tandem stance positions, participants will be asked to place their non-dominant foot behind the dominant foot. For standing on one foot, they will use their non-dominant leg. Participants will be allowed to hold on to wall when changing positions. An investigator will use a stop watch to time each test.
Change of the dynamic posture test for people with osteoporosis from baseline to 3 months | This test will be performed at baseline and within a week after the completion of the intervention
  This test assesses if individuals with osteoporosis hold good posture with two activities. The first, an investigator will observe if participants twist or bend their spines with sit-to-stand-to-sit. The next step of the test will be to observe if they twist or bend spine while lifting a box/crate/foot stool from the floor and set it on the kitchen table/ kitchen counter. For the sit-stand-to-sit test, an investigator will see if they scoot forward symmetrically, push up with both arms, and lean forward through their hips without moving their trunk and when they return to sitting they do not twist or bend their trunk to find the chair and bend through their legs as they return to their chair. For the lifting task we will observe that they bend through their legs, turn with their feet to face the counter and keep the load close to them avoiding trunk flexion or rotation. The test is scored using either a 0 for no or a 1 for yes for each of the elements listed above.
Change in the Self-efficacy for Exercise Scale from baseline to 3 months | This scale will be completed at baseline and within a week after the completion of the intervention
  This scale contains nine items. Each item has a 10-point Likert scale response. The higher the score the greater confidence a person has to exercise.
Perceived readiness to exercise item | This item will be completed at baseline only
  This item will be assess a person's perceived readiness to exercise using a 10-point Likert scale. The higher the score the greater perception of readiness to exercise
Change in Falls Efficacy Scale from baseline to 3 months | This scale will be completed at baseline and within a week after the completion of the intervention
  This scale has 9 items. Participants rate their confidence in performing an activity without falling on a 10-point Likert scale. Higher scores indicate greater confidence in not falling when performing activities.
Change in Godin Leisure-Time Physical Activity Questionnaire from baseline to 3 months | This scale will be completed at baseline and within a week after the completion of the intervention
  This scale assesses the number of times an individual engages in mild, moderate and strenuous leisure time physical activity bouts of at least 15-minute duration in a typical week. This is a 4-item self-administered scale.
Demographic questions | These questions will only be asked at baseline
  We will be asking questions related to race and ethnicity, age, height, and weight.
Intervention satisfaction questions | These questions will only be asked post intervention at 3 months
  This survey has 29 items assessing satisfaction of all aspects of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Donald H Lein Jr, PT, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: Undecided
Since this study is a feasibility study, the investigators are not sharing individual participant data at this time. While outcome data is being collected it will be used to determine effect size and to help shape the intervention further.